CLINICAL TRIAL: NCT06405828
Title: Project ACCESS: A Pilot Randomized Controlled Trial of a Navigator Delivered Model to Enhance Access to Supportive Services for Women of Color With Metastatic Breast Cancer
Brief Title: Enhancing Access to Supportive Services for Women of Color With Metastatic Breast Cancer
Acronym: ACCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa Mazor, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Study-21-01250; K08CA267309 (NIH)
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Breast Cancer; Stage IV Breast Cancer AJCC V7
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACCESS Supportive Care (Experimental): Participants randomized to the intervention arm (n=30) will be connected to the navigator to with the ACCESS Supportive care
  Interventions: Behavioral: ACCESS Supportive Care
- Attention Control (Placebo Comparator): Participants randomized to the attention control arm (n=30) will be connected with an unblinded RC .
  Interventions: Behavioral: Phone sessions

INTERVENTIONS:
Behavioral: ACCESS Supportive Care — ACCESS Supportive Care includes:
  1. Coaching sessions: 6 one-hour weekly Community Navigator led supportive and early palliative care health coaching sessions. Sessions will be hybrid (in-person or virtual) per participant preference.
  2. Monthly check-in: Monthly check-ins (~5-10 minutes) about their supportive care and social determinants of health needs over 16 weeks.
  3. Scheduling of outpatient supportive oncology appointment if interested.
  4. Community linkage: Warm hand offs and connection to community resources to enhance access to support groups, educational workshops, and healthy lifestyle services.
  Arms: ACCESS Supportive Care
Behavioral: Phone sessions — 6 weekly phone sessions, approximately 10 minutes in length each, to review breast cancer and supportive and palliative care resources in NYC and online. The 6 weekly phone sessions will include the topics discussed in the intervention arm but will be informational in nature. The phone sessions will be followed by monthly check-ins (~5 minutes) to review and answer questions about the resources for the duration of 16 weeks.
  Arms: Attention Control

SUMMARY:
Black and Latina women experience disparities in supportive and palliative care access and outcomes. The goal of the proposed pilot study is to evaluate the feasibility and acceptability of a community navigator delivered supportive care intervention for historically underserved populations of women with metastatic breast cancer.

DETAILED DESCRIPTION:
Primary Objectives:

1. Establish the feasibility and acceptability of an adapted navigator delivered supportive care model called ACCESS to address supportive care needs for Black and Latina women with Metastatic Breast Cancer.
2. Determine the potential impact of ACCESS on cancer related distress, symptom burden, and utilization of supportive care services.

OUTLINE: Participants (N=60) are randomized to 1 of 2 groups:

GROUP 1/Intervention Group: Participants complete 6 individualized behavioral/educational sessions focused on social determinants of health and supportive care with a trained community navigator followed by monthly phone call check ins for 4 months. Participants complete questionnaires over the phone with a research coordinator at baseline, 6 and 9 months.

GROUP 2/Attention Control group: Participants complete 6 phone calls with a research coordinator focused on supportive care resources followed by monthly phone call check ins for 4 months. Participants complete questionnaires over the phone with a research coordinator at baseline, 6 months and 9 months.

.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age
* English and/or Spanish speaking
* Self-identify as Latina and/or African American/Black
* Ability to understand and the willingness to sign a written informed consent
* Stage IV breast cancer diagnosis, no time component

Exclusion Criteria:

* Moderate to severe cognitive impairment
* receiving inpatient hospice care
* if patients were previously enrolled in Aim 1 and Aim 2
* currently working with a community navigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identify as a woman
Enrollment: 67 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | at 9 months
  Acceptability evaluates if patients accept the intervention through the ability to recruit 60 participants in 1.5 years and a <20% dropout rate at 9 months
Number of participants remaining in study | at 9 months
  Acceptability evaluates if patients accept the intervention through a <20% dropout rate at 9 months
Number of times navigator communicates with oncology team | 9 months
  Integration evaluates if the navigator can communicate with the supportive oncology and medical oncology team at least 80% of the time.
Number of times participants connect to resources | 9 months
  Integration evaluates if at least 80% of patients can connect to community and clinical resources.
Number of visits | 6 months
  Practicality evaluates if the navigator is able to deliver the intervention in person or virtual. Successful practicality benchmarks include > 80% of the visits conducted.
Number of phone calls | 9 months
  Practicality evaluates if the navigator is able to deliver the intervention in person or virtual. Successful practicality benchmarks include >80% of follow up phone calls conducted.
Number of visits conducted according to the ACCESS manual | 9 months
  Fidelity: This is indicated if >80% of the visits are conducted according to the ACCESS manual.
Change in The Impact of Event Scale - Revised (IES-R) scores | Baseline and 9 months
  Cancer-related distress will be measured through the Impact of Event Scale - Revised (IES-R) is a 22-item instrument to assess distress. Each item is scored 0-4, with full scale from 0-22. Higher scores indicate greater severity of symptoms related to distress.
  Efficacy assessed by mean differences at 9 months as compared to baseline.
Change in The Memorial Symptom Assessment Scale (MSAS) | Baseline and 9 months
  Symptom Burden will be measured through the Memorial Symptom Assessment (MSAS) is a 32 item instrument. Each item is scored from 0 to 4 with full scale from 0-128. A higher score indicates a greater level of symptom distress.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Mazor, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Specify Other Mechanism Following publication and any de-identified data and supportive documents can be requested from melissa.mazor@mountsinai.org